CLINICAL TRIAL: NCT05524363
Title: Prospective and Observational Study of HYPE SCS Stems
Brief Title: Assessment of Safety and Performances of HYPE SCS Stem Associated to NOVAE Sunfit TH Acetabular Cup in Hip Arthroplasty
Acronym: 2020-04
Status: Active, not recruiting | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-04-AMELINE_HYPE_SCS
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hip Arthropathy
Keywords: Total Hip Prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Total hip arthroplasty is the preferred treatment for hip disease (primary or secondary osteoarthritis, osteonecrosis, for example) and femoral neck fractures.

HYPE SCS stems are intended to be used for primary total hip arthroplasties to reduce pain and restore joint mobility of the hip.

Clinical data for HYPE SCS available are not deemed sufficient to support performance and benefits claimed on the whole lifetime of the product.

Thus, in order to maintain compliance with the EU regulation (2017/745) relating to medical devices and following MEDDEV 2.7.1.guidelines, SERF has set up post-market clinical follow-ups (PMCF). This PMCF study aims to generate clinical data in order to confirm these performance of HYPE SCS Stem associated to NOVAE Sunfit TH acetabular cup. In the meantime, through complications faced over the entire period of the study, risks related to the implantation of HYPE SCS stems will be assessed at medium term (5 years). It should be noted that this patient cohort reflects the usual medical care of Hospital Center "J. Monod" of Flers.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Patients covered by health insurance system
* Patients requiring a total hip arthroplasty, implanted swith a femoral stem SCS associated to NOVAE Sunfit TH acetabular cup

Exclusion Criteria:

* Patient who expressed opposition to participation in the study and to the use of his personal data
* Patient unable to understand surgeon's instructions and meet follow-ups requirements
* Patient presenting a contraindication indicated in the IFU of both implantsw
* Patient presenting a contraindication to have an X-ray
* Patients implanted with a femoral stem SCS associated to NOVAE Sunfit TH acetabular cup, in context of off-label use

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recruitment of adults patients representing 120 hips operated between 2020 and 2022 (8 patients have been implanted at both hips).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate according to Kaplan-Meier | per operative period to 5 years
  whatever the cause of revision

SECONDARY OUTCOMES:
Patient satisfaction | per operative period to 5 years
  questionnary with a 4 item-scale
Adverse events | per operative period to 5 years
  Type and occurence of adverse events
Functional improvement | per operative period to 5 years
  This information will be documented through patient questionnary Harris Hip Score
Functional improvement | per operative period to 5 years
  This information will be documented through patient questionnary Devane classification
Pain release | per operative period to 5 years
  This information will be documented through patient questionnary : Harris Hip Score

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier " J. Monod ",, Flers-en-Escrebieux, France